CLINICAL TRIAL: NCT07345390
Title: A Multicenter, Double-blind, Placebo-parallel-controlled Phase Ⅱ Clinical Trial to Evaluate the Safety, Efficacy and Pharmacokinetic Characteristics of KR230109 in Patients With Acne Vulgaris
Brief Title: Safety, Efficacy and Pharmacokinetic Characteristics of KR230109 Cream in Facial Acne Vulgaris
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangxi Kvvit Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KR230109-202503
Record Dates: First submitted 2025-12-25; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KR230109 cream 0.025% (Experimental): Participants applied KR230109 cream once daily for 12 consecutive weeks.
  Interventions: Drug: KR230109 cream 0.025%
- KR230109 cream 0.05% (Experimental): Participants applied KR230109 cream once daily for 12 consecutive weeks.
  Interventions: Drug: KR230109 cream 0.05%
- placebo (Placebo Comparator): Participants applied placebo once daily for 12 consecutive weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KR230109 cream 0.025% — KR230109 cream 0.025% is indicated for the topical treatment of acne vulgaris in patients
  Arms: KR230109 cream 0.025%
Drug: KR230109 cream 0.05% — KR230109 cream 0.05% is indicated for the topical treatment of acne vulgaris in patients
  Arms: KR230109 cream 0.05%
Drug: Placebo — Vehicle cream manufactured to mimic look and feel of KR230109 Cream but without the active ingredient.
  Other Names: Vehicle cream
  Arms: placebo

SUMMARY:
This study will evaluate the safety, efficacy and pharmacokinetics of KR230109 cream compared with placebo in Patients (18-40 Years) with Acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 40 years old (as of the time of signing the informed consent form), regardless of gender;
2. Patients clinically diagnosed with mild to moderate facial acne vulgaris (refer to the "Chinese Acne Treatment Guidelines" 2019 revised edition), and with an overall facial IGA (Investigator Global Assessment) score of 2 to 3 by the study doctor;
3. Baseline requirements: For patients with mild to moderate acne, the count of facial inflammatory lesions (papules and/or pustules) should be >=10 and <=40; the count of non-inflammatory lesions (open and/or closed comedones) should be >=20 and <=60; no facial nodules should exist;
4. Participants must be willing to use only non-acne-treating skin care products during the trial and comply with the precautions required by the protocol;
5. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the written informed consent form, and be able to complete the entire trial process as required;
6. From the time of signing the informed consent form to 3 months after the last administration, female participants of childbearing age or male participants whose partners are of childbearing age must agree and be able to take effective contraceptive measures, such as avoiding sexual activity or using reliable contraceptive methods like condoms or intrauterine devices.

Exclusion Criteria:

1. Those known to be allergic to KR230109 or drugs with the same mechanism of action such as tazarotene, adapalene, or any of their components;
2. Those with a history of any serious clinical systemic diseases or surgeries, such as diseases of the circulatory system, nervous system, hematological system, immune system, or mental system;
3. Those with concurrent other obvious skin diseases at the affected area that may affect the clinical evaluation of the researchers or require concurrent treatment, such as solar dermatitis, psoriasis, seborrheic dermatitis, rosacea, eczema, severe acne, and extremely severe acne (such as conglobate acne, fulminant acne, etc.);
4. Those with secondary acne, such as occupational acne and acne caused by corticosteroids;
5. Those with facial skin or hair conditions that may interfere with clinical assessment (such as significant beards, sideburns, or mustaches);
6. Those who plan to use any adjunctive therapies or concomitant treatments for acne during the trial;
7. Those who have used acne-specific functional skin care products within one week before the start of treatment;
8. Those who have used topical retinoids, antibiotics, corticosteroids, or other topical acne treatments on the face within two weeks before the trial;
9. Those who have taken oral retinoids, antibiotics, corticosteroids (including intramuscular or intralesional injections, except for stable use of inhaled, intranasal, or intraocular corticosteroids for the treatment of underlying diseases and without impact on acne treatment), spironolactone, or other acne medications within four weeks before the trial;
10. Those who have undergone physical or chemical acne treatments within four weeks before the trial;
11. Those who have participated in other clinical trials and used trial drugs or medical devices within 90 days before screening or plan to participate in other clinical trials during the trial;
12. Those whose vital signs, physical examinations, laboratory tests (blood routine, urine routine, blood biochemistry), electrocardiograms, etc., are abnormal and have clinical significance as assessed by the researchers and may affect the evaluation of this trial;
13. Those who are positive for hepatitis B surface antigen, hepatitis C antibody, syphilis-specific antibody, or human immunodeficiency virus antibody;
14. Pregnant or lactating women or those with positive blood or urine pregnancy tests;
15. Those who need prolonged or excessive exposure to sunlight, such as sunbathing;
16. Those with a history of alcohol abuse or drug abuse;
17. Those who, in the opinion of the researchers, have poor compliance, or have conditions that may interfere with the study outcome, or those who, in the opinion of the researchers, have any other conditions that make them unsuitable for participation in this clinical trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The percentage change from baseline in the count of non-inflammatory facial lesions | week 12
  The percentage change from baseline in the count of non-inflammatory facial lesions at Week 12 compared with placebo in each treatment group.
The percentage change from baseline in the count of inflammatory facial lesions | week 12
  The percentage change from baseline in the count of inflammatory facial lesions at Week 12 compared with placebo in each treatment group.

SECONDARY OUTCOMES:
The average percentage change from baseline in the counts of inflammatory and non-inflammatory skin lesions | week 2,4,8
  The average percentage change from baseline in the counts of inflammatory and non-inflammatory skin lesions at weeks 2, 4, 8 of treatment compared with placebo for each treatment group.
The absolute change from baseline in the counts of inflammatory and non-inflammatory skin lesions | week 2,4,8,12
  The absolute change from baseline in the counts of inflammatory and non-inflammatory skin lesions at weeks 2, 4, 8, 12 of treatment compared with placebo for each treatment group.
The average percentage change and absolute change from baseline in the total skin lesion count | week 2,4,8,12
  The average percentage change and absolute change from baseline in the total skin lesion count at weeks 2, 4, 8, 12 of treatment compared with placebo for each treatment group.
The proportion of participants in each treatment group with at least a 2-point reduction in IGA score from baseline and an IGA score of 0 or 1 | week 2,4,8,12
  The proportion of participants in each treatment group with at least a 2-point reduction in IGA score from baseline and an IGA score of 0 or 1 at weeks 2, 4, 8, 12 of treatment compared with placebo.
Safety endpoints | from day 1 to week 12
  Adverse events (AEs), local skin reactions (LSRs), physical examinations, vital signs, electrocardiograms (ECGs), and abnormal clinical laboratory tests (blood routine, blood biochemistry, urine routine).
Steady-state PK parameters of KR230109: Cmax,ss. | week 4
  Steady-state PK parameters of KR230109: Cmax,ss.
Steady-state PK parameters of KR230109: AUC0-24h,ss, etc. | weeks 4
  Steady-state PK parameters of KR230109: AUC0-24h,ss, etc.